CLINICAL TRIAL: NCT02694874
Title: Rosiglitazone Adjunctive Therapy for Severe Malaria in Children
Acronym: ROSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: University Health Network, Toronto (Other); Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROSI_v03_22072015
Record Dates: First submitted 2015-12-09; First posted 2016-03-01 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Malaria
Keywords: Adjunctive treatment; Severe malaria
MeSH Terms: conditions — Malaria | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone (Experimental): Participants will receive rosiglitazone 0.045mg/kg/dose twice daily dosing, for 4 days
  Interventions: Drug: Rosiglitazone
- Placebo (Placebo Comparator): Participants will receive placebo (grounded placebo powder) at a dose of 0.045mg/kg/dose twice daily for 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — This is the experimental drug, rosiglitazone, being tested against placebo to assess its efficacy as an adjunctive treatment for severe malaria
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Placebo — This is the placebo control
  Other Names: crushed powder placebo
  Arms: Placebo

SUMMARY:
Even with optimal anti-malaria therapy and supportive care, severe and cerebral malaria are associated with a 10-30% mortality rate and neurocognitive deficits in up to 33% of survivors. Adjunctive therapies that modify host immune-pathological processes may further improve outcome over that possible with anti-malarials alone. Investigators aim to evaluate a PPARγ agonist ( "rosiglitazone") as adjunctive therapy for severe malaria.

DETAILED DESCRIPTION:
Although the use of artemisinin-based therapy has improved outcomes in severe malaria, the mortality rates remain high. Adjunctive therapies that target the underlying immunopathology may further reduce morbidity and mortality in severe and cerebral malaria beyond that possible with anti-malarials alone. Pre-clinical data have established a beneficial role for PPARγ agonists in experimental cerebral malaria. A proof-of-concept randomized clinical trial of uncomplicated malaria in Thailand has extended these findings to an informative patient population, showing that adjunctive treatment with the PPARγ agonist rosiglitazone improves parasite clearance, and reduces biomarkers of inflammation (IL-6 and MCP-1) and endothelial activation (Ang-2 to Ang-1 ratio), and increases neuro-protective pathways (BDNF). The previous clinical trial also established the safety and tolerability of short course rosiglitazone in adults with malaria infection. Importantly, rosiglitazone does not induce insulin release or hypoglycemia in malaria-infected patients. Based on these data, and on studies demonstrating neuro-protective effects on PPARγ agonists in CNS disease and injury, the investigators believe that PPARγ agonists are promising candidates for adjunctive therapy for severe and cerebral malaria.

In this study the efficacy of rosiglitazone vs. placebo control as adjunct to standard of care anti-malarial therapy in children with severe (including cerebral) malaria will be tested.

The underlying hypothesis is that the addition of rosiglitazone to standard antimalarial therapy in severe P. falciparum infection is safe and will result in improved clinical outcomes and lower rates of long-term neurocognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-12 years
* Positive 3-band (HRPII plus pLDH) P. falciparum rapid diagnostic test (RDT) and microscopy confirmed malaria infection with parasitemia >2500 parasites/microlitre if microscopy is available in a timely manner at the time of randomization.
* One or more features of severe malaria: repeated seizures (two or more generalized seizures in 24 h); prostration (in children 1 year and older, the child is unable to sit unsupported or stand although was able to before the illness); impaired consciousness (Blantyre Coma Score <5 in children 1 to 4 years, GCS <14 for children ≥ 5 years); respiratory distress: age related tachypnea with sustained nasal flaring, deep breathing or subcostal retractions
* Requiring hospitalization and parenteral artesunate for their malaria infection based on admitting physician assessment

Exclusion Criteria:

* P. falciparum RDT negative OR infection not confirmed by light microscopy or not reaching the predefined inclusion criterion parasitemia threshold according to age
* Uncomplicated malaria infection not requiring hospitalization
* Presenting with severe malaria anemia (SMA) alone (Hb < 50g/L)
* Known underlying illness: neurological or neurodegenerative disorders, cardiac, renal, or hepatic disease, diabetes, epilepsy, cerebral palsy, children known to be HIV-1 positive and receiving antiretroviral treatment*
* Previous treatment with a TZD
* Unable to remain in research site region for the follow up period

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change in serum Ang-2 levels in the first 96 hours of hospital admission. | first 96 hours of hospital admission.
  We will assess the effect of the intervention (vs. placebo) on Ang-2 levels as a biomarker of severe disease in severe malaria

SECONDARY OUTCOMES:
Time to clinical recovery | up to 96 hours after hospital admission
  Time to recovery including:
  1. Time to fever resolution for at least 24h. Temperature measurements will be taken at admission and every 4h for the first 4 days, and then every 12h until 2 normal results (<37.5oC) are reported.
  2. Time to sit unsupported
  3. Time to hospital discharge
Time to parasitological recovery | up to 96 hours after hospital admission
  Time to parasitological recovery: Time (in hours) to clearance of parasitemia from the blood (both 50% and 90% decrease from admission baseline value). Parasitemia will be quantified at admission and every 6h, for 4 days or until 2 negative readings are reported.
Mortality | first 48h post-hospital admission and at 14 days post-hospital admission
  Mortality in the first 48h post-hospital admission and at 14 days post-hospital admission
Blood lactate levels, assessed at admission, every 12h for 24 hours then daily for Blood lactate levels | Assessed at admission, every 12h for 24 hours then daily for 4 days, and once on day 14 and 6 month follow ups
  Blood lactate levels, assessed at admission, every 12h for 24 hours then daily for 4 days, and once on day 14 and 6 month follow ups
Change in levels of biomarkers of host response | at admission, every 12h for 24 hours then daily for 4 days, and once on day 14 and 6 month follow ups
  Change in levels of biomarkers of host response at admission, every 12h for 24 hours then daily for 4 days, and once on day 14 and 6 month follow ups
Blood glucose levels | up to 96 hours after hospital admission
  Blood glucose levels assessed at admission and every 6h for the first 48h, and then every 24h for following 2 days
Cardiac effects | from baseline to 24h, and day 4
  Monitor for cardiac effects by conducting ECG at baseline, at 24h (immediately before third doses of rosiglitazone and artesunate treatment are administered) and at the end of rosiglitazone treatment (day 4). Main outcome of interest will be changes in QTc from baseline to the two different time points.
Biochemical and hematological parameters | up to 96 hours after hospital admission
  Biochemical and hematological parameters including: AST, ALT, creatinine, complete blood count (e.g. hemoglobin, WBC and differential, hematocrit, platelet count) will be assessed at admission and every 24h until day 4
AE/SAE | up to day 14 after hospital admission
  AE/SAE monitored using the pediatric toxicity tables modified from the US National Institutes of Allergy and Infectious Diseases
Neurocognitive outcomes | From baseline to 6 months post discharge, and 18 months post discharge
  Participants with Adverse Events that Are Related and unrelated to Treatment by a variety of standard neurocognitive tests

CONTACTS AND LOCATIONS:
Overall Officials: Eusebio Macete, PhD, Study Director — Fundaçao Manhiça
Locations (1):
- Centro de Investigação em Saude da Manhiça, Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Varo R, Crowley VM, Mucasse H, Sitoe A, Bramugy J, Serghides L, Weckman AM, Erice C, Bila R, Vitorino P, Mucasse C, Valente M, Ajanovic S, Balanza N, Zhong K, Derpsch Y, Gladstone M, Mayor A, Bassat Q, Kain KC. Adjunctive rosiglitazone treatment for severe pediatric malaria: A randomized placebo-controlled trial in Mozambican children. Int J Infect Dis. 2024 Feb;139:34-40. doi: 10.1016/j.ijid.2023.11.031. Epub 2023 Nov 25. PMID 38013152
- [Derived] Varo R, Crowley VM, Sitoe A, Madrid L, Serghides L, Bila R, Mucavele H, Mayor A, Bassat Q, Kain KC. Safety and tolerability of adjunctive rosiglitazone treatment for children with uncomplicated malaria. Malar J. 2017 May 23;16(1):215. doi: 10.1186/s12936-017-1858-0. PMID 28535809